CLINICAL TRIAL: NCT04020068
Title: Diabetes Cohort in French Amazonia
Acronym: CoDiAm
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier de Cayenne (Other)
Responsible Party: Sponsor
Other Study IDs: CODIAM
Record Dates: First submitted 2019-07-10; First posted 2019-07-15 (Actual); Last update posted 2019-07-15 (Actual); Status verified 2019-07

CONDITIONS: Diabetes Mellitus; Adults
Keywords: Diabete; French Guiana
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples Without DNA — blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
CoDiAm aims to collect clinical, biological and social data of diabetic patients in French Guiana.

DETAILED DESCRIPTION:
Diabetes is a very common disease in French Guiana. This disease is caused by the body's inability to metabolise sugar properly. A diet and treatment with tablets are enough for some patients, while others may need insulin injections. In the long term, high blood sugar levels may cause problems to the small and large blood vessels in the body. This is complicated by nerve, renal and retinal damage, as well as increased risks of cardiac and vascular events (such as strokes or heart attacks.) It appears that diabetes is more common and more severe in French Guiana than in other parts of France. It seems that the types of diabetes found here are more variable than those found in France, and that patients tend to be diagnosed at a later stage. We would this like to better understand diabetes and its evolution in French Guiana.

This research is aimed at diabetic patients and it is being carried out in the Andrée Rosemon Hospital Centre, the Ouest Guyanais Hospital Centre as well as in other Primary Healthcare Centres. At some point in the future, some private health centres may also invite their patients to take part in this study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diabetes
* At least 18 years old

Exclusion Criteria:

* Less than 18 years old
* Patients under legal guardianship
* Patients' refusal to participate
* Patients living outside French Guiana

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diabetic patients living in French Guiana
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2019-04-08 (Actual); Primary Completion 2021-04-08 (Estimated); Study Completion 2021-05-08 (Estimated)

PRIMARY OUTCOMES:
Improvement of patient care | 2 years
  Number of health complications in diabetes mellitus ...

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier de Cayenne, Cayenne, French Guiana, France

IPD SHARING:
Plan to Share IPD: No